CLINICAL TRIAL: NCT05370781
Title: Michigan Men's Diabetes Project 2
Acronym: MenD 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jaclynn Hawkins, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00200469
Record Dates: First submitted 2022-05-03; First posted 2022-05-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer led diabetes self-management support (PLDSMS) (Experimental): Participants in the PLDSMS arm will receive 10 hours of diabetes self-management education (DSME) with a certified diabetes care and education specialist. This group will then transition into monthly 90-minute diabetes self-management support (DSMS) with trained peer leaders for 6 months. After the DSMS sessions, the group will transition into 6 months of ongoing support and will be encouraged to continue DSMS through initiatives that are important to them.
  Interventions: Behavioral: Peer Led Diabetes Self-Management Support; Behavioral: Diabetes Self-Management Education
- Control Group (Active Comparator): Participants in the control group will receive 10 hours of diabetes self-management education (DSME) with a certified diabetes care and education specialist.
  Interventions: Behavioral: Diabetes Self-Management Education

INTERVENTIONS:
Behavioral: Peer Led Diabetes Self-Management Support — While the effectiveness of peer-led interventions delivering diabetes-related education and support for short-term clinical, psychosocial, and behavioral improvements is well-established, older Black men in particular are less likely to participate and are at a higher risk of drop-out from these studies. This intervention aims to determine if using older Black men as peer leaders to other older Black men will improve retention rates for this population.
  Arms: Peer led diabetes self-management support (PLDSMS)
Behavioral: Diabetes Self-Management Education — Participants will attend 10 hours of virtual group diabetes self-management education classes led by a certified diabetes care and education specialist through the online HIPPA compliant Zoom platform.

SUMMARY:
The Michigan Men's Diabetes Project 2 (MenD 2) is an 18-month pilot randomized clinical trial. We are looking to recruit 60 Black men with type 2 diabetes (need to have diagnosis for at least 6 months) that are over the age of 21. Interested participants need to be under the care of a physician for their diabetes, have access to reliable transportation for study activities, and be willing to participate in 4 health assessments where they will get their A1C, blood pressure, height, and weight measured and they will complete a survey. All participants will receive 10 hours of diabetes self-management education with a Certified Diabetes Care and Education Specialist. Participants randomized to the intervention arm will also be offered 6 months of monthly diabetes self-management support (DSMS) sessions with trained Peer Leaders who are also Black men with type 2 diabetes. After the 6 months of support, this group will transition into 6 months of ongoing support where they can continue DSMS and/or other diabetes related initiatives that are important to the group and chosen by the group. Due to the COVID-19 pandemic, DSME and DSMS sessions will likely be held via Zoom, ongoing support sessions have potential to be in person. The 4 health assessments will take place at baseline, 3-months, 9-months, and 15-months.

ELIGIBILITY:
Inclusion Criteria:

* Black/African American males, age 21 years or older with diagnosis of T2D for six months, transportation to attend program activities, under the care of a physician for diabetes, and willing to attend group delivered sessions.

Exclusion Criteria:

* We considered restricting eligibility to a higher-risk population of participants with A1c ≥ 8%. Preliminary data suggest that over 50% of the proposed study sample will have an A1c ≥ 8%. Focusing on all older Black men with T2D allows us to cast a wide net for secondary prevention and public health impact.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation of gender identity
Enrollment: 48 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | baseline, 3-months, 9-months, 15-months
  Anthropometric/clinical data
Change in Regimen Adherence | baseline, 3-months, 9-months, 15-months
  Survey data

SECONDARY OUTCOMES:
Change in Depression | baseline, 3-months, 9-months, 15-months
  survey data
Change in Body Mass Index | baseline, 3-months, 9-months, 15-months
  Anthropometric data/clinical data
Change in Blood Pressure | baseline, 3-months, 9-months, 15-months
  Anthropometric data/clinical data
Change in Diabetes Social Support | baseline, 3-months, 9-months, 15-months
  survey data
Change in Diabetes-Related Distress | baseline, 3-months, 9-months, 15-months
  survey data
Change in Diabetes Quality of Life | baseline, 3-months, 9-months, 15-months
  survey data
Change in Adherence to gender norms | baseline, 3-months, 9-months, 15-months
  survey data

CONTACTS AND LOCATIONS:
Overall Officials: Jaclynn Hawkins, PhD, Principal Investigator — University of Michigan, School of Social Work
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Hawkins J, Sengupta S, Kloss K, Kurnick K, Ewen A, Nwawkwo R, Funnell M, Mitchell J, Jones L, Piatt G. Michigan men's diabetes project II: Protocol for peer-led diabetes self-management education and long-term support in Black men. PLoS One. 2023 Mar 2;18(3):e0277733. doi: 10.1371/journal.pone.0277733. eCollection 2023. PMID 36862648

DOCUMENTS (2):
  • Informed Consent Form: Participant Consent Form (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT05370781/ICF_000.pdf
  • Informed Consent Form: Peer Leader Consent Form (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT05370781/ICF_001.pdf